CLINICAL TRIAL: NCT03729934
Title: Effects of Ketones Supplementation on Postprandial Lipemia
Brief Title: Ketones Supplementation and Postprandial Lipemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Dissertation for student changed.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Eric P. Plaisance, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KBS2018
Record Dates: First submitted 2018-10-23; First posted 2018-11-05 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Overweight and Obesity; Overweight; Triglycerides High
MeSH Terms: conditions — Obesity; Overweight; Hypertriglyceridemia | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): This arm receives no treatment control.
- Ketone Ester (Experimental): This arm receives 25 g ketone ester.
  Interventions: Dietary Supplement: Ketone Ester
- Ketone Salt (Experimental): This arm receives 25 g ketone salt.
  Interventions: Dietary Supplement: Ketone Salt

INTERVENTIONS:
Dietary Supplement: Ketone Ester — This arm receives 25 g ketone ester.
  Arms: Ketone Ester
Dietary Supplement: Ketone Salt — This arm receives 25 g ketone salt.
  Arms: Ketone Salt

SUMMARY:
This study determines whether different forms of ketones supplemented prior to a meal lower the triglyceride (fat) content in the blood of overweight and obese individuals. Through a randomized crossover design, participants (n=15) will participate in each of the following three experimental groups (no treatment control, ketone ester, ketone salt), with a 5-14 day washout period between each experimental visit.

DETAILED DESCRIPTION:
Previous studies conducted by the investigative team in rodents show that male mice fed a diet containing 30% ketone ester (by kcals) results in greater fecal content and energy loss. While the investigators are unsure of the exact macronutrient content of the energy loss, the hypothesis is that the energy excretion is attributed to lower fat absorption. In the context of this study, it's hypothesized that ketone salts and ketone esters (both available commercially and used for a variety of health-related claims) will reduce the absorption of dietary fats leading to lower circulating triglyceride concentrations if consumed prior to a high-fat mixed meal. If the hypothesis is correct, ketones supplementation could become a valuable strategy to reduce the rise in circulating triglycerides often present in obesity. Triglyceride concentrations in the blood following a meal have been linked to development of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese men as defined by a BMI of greater than or equal to 25 kg/m2, but less than 35 kg/m2
* Between the ages of 25 and 45 years
* Fasting triglyceride levels less than 250 mg/dL

Exclusion Criteria:

* Participates in regular physical activity (≥3 days/week at 30 minutes or more per day)
* Diagnosed cardiovascular disease or metabolic disease (type 1 or type 2 diabetes)
* Currently following a low carbohydrate (<100 g/day) diet
* Lost greater than or equal to 5% body weight over the last 2 months
* Alcohol/smoking/antibiotics

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline plasma glucagon-like peptide 1 at 240 minutes | 0, 30, 60, 120, 180, and 240 minutes post-supplement consumption
  Plasma levels of glucagon-like peptide 1 in pg/L
Change from baseline serum triglycerides at 240 minutes | 0, 30, 60, 120, 180, and 240 minutes post-supplement consumption
  Serum levels of triglycerides in mg/DL
Change from baseline serum glucose at 240 minutes | 0, 30, 60, 120, 180, and 240 minutes post-supplement consumption
  Serum levels of glucose in mg/dL
Change from baseline serum Insulin at 240 minutes | 0, 30, 60, 120, 180, and 240 minutes post-supplement consumption
  Serum levels of insulin in pmol/L
Change from baseline serum B-hydroxybutyrate at 240 minutes | 0, 30, 60, 120, 180, and 240 minutes post-supplement consumption
  Serum levels of B-hydroxybutyrate in mmol/L
Change from baseline plasma ghrelin at 240 minutes | 0, 30, 60, 120, 180, and 240 minutes post-supplement consumption
  Plasma levels of ghrelin in pg/mL
Change from baseline plasma leptin at 240 minutes | 0, 30, 60, 120, 180, and 240 minutes post-supplement consumption
  Plasma levels of leptin in ng/mL